CLINICAL TRIAL: NCT06889506
Title: Assessment of Interleukin-4 Tissue and Serum Levels in Pityriasis Lichenoides Chronica Patients : a Case- Control Study
Brief Title: Interleukin-4 in Pityriasis Lichenoides Chronica
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Mona Mostafa Korany Mahmoud, principal investigator, Cairo University
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: Dermatology 20
Record Dates: First submitted 2025-03-16; First posted 2025-03-21 (Actual); Last update posted 2025-03-21 (Actual); Status verified 2025-01

CONDITIONS: Pityriasis Lichenoides
MeSH Terms: conditions — Pityriasis Lichenoides

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- PLC patients (Active Comparator): one skin biopsy (lesional) and serum sample will be taken from every patient
  Interventions: Procedure: skin biopsy and serum sample
- healthy controls (Experimental): a skin biopsy and serum sample will be taken from each control sample
  Interventions: Procedure: skin biopsy and serum sample

INTERVENTIONS:
Procedure: skin biopsy and serum sample — skin biopsy from lesional skin and serum sample will be taken from each patient . also a skin biopsy and serum sample will be taken from each healthy control

SUMMARY:
assessment of the level of interleukin 4 (IL-4) in the lesional skin and serum of PLC patients and compare its level with healthy controls.

DETAILED DESCRIPTION:
measuring the level of Interleukin 4 in lesional skin and it's serum level using ELIZA in patients with Pityriasis lichenoides chronica and comparing the levels with healthy controls levels

ELIGIBILITY:
Inclusion Criteria:

* Patients with pityriasis lichenoides Chronica (PLC): either with the classical presentation papular or hypo-pigmented macules and patches that proved histopathologically to be PLC.
* Both genders
* Age group ≥ 8 years

Exclusion Criteria:

* Patients with other skin diseases
* Patient received treatment for PLC within period less than three months
* Pregnant patients
* Lactating patients

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2025-04-01 (Estimated); Primary Completion 2025-07 (Estimated); Study Completion 2025-07 (Estimated)

PRIMARY OUTCOMES:
Assessment of tissue and serum levels of interleukin 4 (IL -4) in pityriasis lichenoides chronica (PLC) patients and normal controls. | 6 months
  measurement of tisssue and serum levels of interleukin 4 (IL -4) in pityriasis lichenoides chronica (PLC) patients and comparing them with normal controls to control and verify the hypothesisof involvement of IL-4 in the pathogenesis of PLC